CLINICAL TRIAL: NCT01413464
Title: The Risk of Thromboembolism in Patients Post Renal Transplantation (REPORT) Study
Brief Title: The Risk of Venous Clotting in Patients After Renal Transplant
Acronym: REPORT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Christine Ribic, Nephrologist, St. Joseph's Healthcare Hamilton
Other Study IDs: 10-3440
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Venous Thrombosis; End Stage Renal Failure With Renal Transplant; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Renal Transplant; Venous Thrombosis; Deep Vein Thrombosis; Prophylaxis; Bleeding
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples from participants are being banked at various timepoints.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clots that develop in the deep veins of the legs or the lungs can result in pain, heart and lung disease and may lead to death if unrecognized or not treated. Risk factors for developing clots include surgery, hospitalization and/or being immobile. Up to 10 to 40% of people may develop a clot during or after their hospital stay or surgery, and sometimes these clots do not cause symptoms. In order to help reduce the risk of developing a clot in the legs or lungs, many people undergoing surgery receive a small dose of a blood thinner in hospital after their surgery is completed. Although prescription of a low dose blood thinner is routine practice after most surgeries, the risk or benefit of blood thinners after kidney transplant surgery is still not clear. Given this, many transplant physicians differ in prescribing practices of low dose blood thinners after kidney transplant surgery. More information is needed about the risk of clotting and bleeding in people after kidney transplant surgery so that physicians can become more unified in deciding whether a low dose blood thinner would protect patients after kidney transplant without producing harm.

The REPORT study is designed to examine the risk of clotting in the legs or lungs in people after kidney transplant surgery as well as the risk of bleeding. Ultrasounds of the legs will be performed at various time points after surgery for up to one year to screen for blood clots. People participating in this study will also be screened and monitored for bleeding after surgery. Although this study will also examine the prescription practices of physicians, no blood thinners will be given or withheld from participants as a result of this study. Physicians will prescribe blood thinners as per their usual practice after kidney transplant. Overall, the goal of the study is to find out how frequent clotting and/or bleeding is after kidney transplant surgery, which will help in making recommendations regarding the use of low dose blood thinners in people after their surgery.

Ultrasound scanning of the legs is a safe test that does not cause physical pain and has no risk of causing injury. Participation in this study will provide the benefit of additional monitoring with several ultrasound tests after surgery, screening for clots in the legs which can cause health risks and even death if unrecognized. If a clot is found, it will be treated promptly and according to current medical standards under the care of a specialist.

In the long term, the results of this study will help improve health care delivery to people undergoing kidney transplant with the goal of decreasing potential complications such as clotting and/or bleeding. Currently, there are no guidelines available to guide physician's in the use of a low dose blood thinner after kidney transplant surgery. This study will help determine the risk of clotting or bleeding and help us make recommendations that will reduce potential risks and complications for people undergoing kidney transplant in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age admitted to St. Joseph's Healthcare Hamilton for renal transplantation.

Exclusion Criteria:

* Patients requiring therapeutic and/or bridging anticoagulation pre and post operatively.

Patients requiring therapeutic anticoagulation preoperatively and anticipate therapeutic anticoagulation postoperatively within 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to St. Joseph's Healthcare Hamilton (McMaster University affiliated teaching hospital) to the Renal Transplant Ward for renal transplantation.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Deep Vein Thrombosis or Pulmonary Embolism | 12 months
  Venous thromboembolism (deep vein thrombosis and pulmonary embolism) is screened for at regular study intervals for 12 months and upon clinical suspicion of an event.

SECONDARY OUTCOMES:
Bleeding | 12 months
  Clinically significant bleeding is collected with subjective measures and is adjudicated.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada